CLINICAL TRIAL: NCT03434535
Title: A Pilot Study of Remote Monitoring to Improve Health Related Quality of Life of Men Following Prostate Cancer Treatment.
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Johns Hopkins University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Other
Other Study IDs: IRB00156374
Record Dates: First submitted 2018-02-06; First posted 2018-02-15 (Actual); Last update posted 2019-12-13 (Actual); Status verified 2019-12

CONDITIONS: Health-Related Quality Of Life

STUDY DESIGN:
Who Masked: Participant
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Intervention (Experimental): The participants will complete a digital health-related quality of life survey on a programmed tablet at baseline and each month for the following 3-6 months. They will also receive an activity sensor and weight scale. Health state data from this group will be generated over a 3-6 month period and remotely monitored. These data will be used to provide personalized feedback regarding the participant's progress towards established goals.
  Interventions: Device: Technology Intervention
- Control (No Intervention): The participants will complete a digital health-related quality of life survey on a programmed tablet at baseline and each month for the following 3-6 months.

INTERVENTIONS:
Device: Technology Intervention — A combination of existing technology and a new app developed by InHealth Measurement Corp to (1) remotely monitor a participant's activity level and weight and (2) remotely provide updates to the participants regarding their progress towards the goals established in the Prostate Cancer Foundation Health and Wellness guidelines.
  Other Names: Fitbit Alta HR; Fitbit Aria
  Arms: Intervention

SUMMARY:
The purpose of this study is to determine the feasibility of using digital technology and remote monitoring to track health-related measures in men following prostate cancer treatment. Half of the participants will receive tools to monitor their activity and weight, as well as personalized feedback on these measures, while the other half will receive standard of care. Health related quality of life measure will be collected from both groups.

DETAILED DESCRIPTION:
The purpose of this study is to determine the feasibility of using digital technology and remote monitoring to track health-related measures in men following prostate cancer treatment. All participants will complete a health-related quality of life survey each month for 3 months. The digital survey will be administered on a programmed tablet. The participants in the intervention group will also receive an activity sensor and weight scale. Health state data from this group will be generated over a 3-6 month period and remotely monitored. These data will be used to provide personalized feedback regarding the participant's progress towards established goals. Health-related quality of life will be compared between participants in the intervention group, who receive (1) tools to monitor their activity and weight and (2) personalized feedback, versus participants in the control group, who receive standard of care. The potential improved adherence to healthy behaviors of the participants receiving personalized feedback may translate to to improved health-related quality of life.

ELIGIBILITY:
Inclusion Criteria:

* Participants must have localized prostate cancer.
* Participants must have received treatment at Johns Hopkins
* Participants must be classified as overweight (body mass index ≥ 25).
* Participants must have wi-fi in their homes.

Exclusion Criteria:

* Anyone who is unable to give informed consent will be excluded
* Anyone who is physically unable to participate in physical activity will be excluded.

Sex: Male | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 9 (Actual)
Dates: Start 2018-07-11 (Actual); Primary Completion 2019-10-16 (Actual); Study Completion 2019-10-16 (Actual)

PRIMARY OUTCOMES:
Health-Related Quality of Life | Baseline
  36-Item Short Form (SF) Survey. This survey is a patient-reported survey of patient health. The SF-36 consists of eight scaled scores, which are the weighted sums of the questions in their section and the scores range from 0-100. A score of 0 is equivalent to maximum disability and a score of 100 is equivalent to no disability.
Health-Related Quality of Life | 1 month after baseline
  36-Item Short Form Survey. This survey is a patient-reported survey of patient health. The SF-36 consists of eight scaled scores, which are the weighted sums of the questions in their section and the scores range from 0-100. A score of 0 is equivalent to maximum disability and a score of 100 is equivalent to no disability.
Health-Related Quality of Life | 2 months after baseline
  36-Item Short Form Survey. This survey is a patient-reported survey of patient health. The SF-36 consists of eight scaled scores, which are the weighted sums of the questions in their section and the scores range from 0-100. A score of 0 is equivalent to maximum disability and a score of 100 is equivalent to no disability.
Health-Related Quality of Life | 3 months after baseline
  36-Item Short Form Survey. This survey is a patient-reported survey of patient health. The SF-36 consists of eight scaled scores, which are the weighted sums of the questions in their section and the scores range from 0-100. A score of 0 is equivalent to maximum disability and a score of 100 is equivalent to no disability.

CONTACTS AND LOCATIONS:
Overall Officials: Peter Searson, PhD, Principal Investigator — Johns Hopkins University
Locations (1):
- Johns Hopkins Hospital, Baltimore, Maryland, United States